CLINICAL TRIAL: NCT01268241
Title: International Observational Retrospective Case Review of Efficacy and Safety of Switch Between Agalsidase Beta to Agalsidase Alfa for Enzyme Replacement in Males and Females With Anderson-Fabry Disease
Brief Title: The Efficacy and Safety of Switch Between Agalsidase Beta to Agalsidase Alfa for Enzyme Replacement in Patients With Anderson-Fabry Disease
Acronym: SWITCH
Status: Completed | Type: Observational
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: SW02/2010
Record Dates: First submitted 2010-12-28; First posted 2010-12-29 (Estimated); Last update posted 2021-04-09 (Actual); Status verified 2020-04

CONDITIONS: Fabry Disease; Fabry´s Disease; Anderson-Fabry Disease
Keywords: Fabry Disease; Fabry´s Disease; Anderson-Fabry Disease
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Plasma and urine GB3 and lyso-GB3 and agalsidase antibodies will be analyzed in central laboratories, there is consent for extra blood samples to be taken (at the time of the switch and after 6, 12 and 24 months)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observation: Hemizygous male or heterozygous female patients of any age with genetically confirmed diagnosis of Anderson-Fabry disease.

SUMMARY:
The current approved treatment for Fabry disease is enzyme replacement therapy (ERT). There are actually 2 products in this therapeutic class available: Replagal® (agalsidase alfa) and Fabrazyme® (agalsidase beta). Both are indicated for long-term treatment in patients with a confirmed diagnosis of Fabry disease (alfa-galactosidase A deficiency). Both have been commercially available in Europe for almost 10 years, yet little information is available about the clinical and safety profile of patients who switch from one therapy to the other. An extended shortage of Fabrazyme® that began in June 2009 has necessitated that a large number of patients switch from Fabrazyme® to Replagal®. This offers the possibility to study the clinical status and adverse events in patients who switch from Fabrazyme® to Replagal® on a large-scale basis. In addition, as a result of the increasing Fabrazyme® shortage, many of these patients received a reduced dosage of Fabrazyme® for an extended period before transitioning to treatment with Replagal®.

DETAILED DESCRIPTION:
Aim:

Anderson-Fabry disease is an X-linked lysosomal storage disorder resulting from deficiency of the hydrolytic enzyme alfa galactosidase A. Trials of specific therapy by replacement of alfa galactosidase A were commenced in 1999 and subsequently two preparations of alfa galactosidase A received marketing approval by the EMEA in 2001. Clinical trials, observational studies and registry data have provided evidence for efficacy of enzyme replacement therapy (ERT) with alfa galactosidase A in improving symptoms of pain, gastrointestinal disturbance, hypohidrosis, left ventricular mass index, glomerular filtration rate and quality of life in men. There is currently no long-term data showing the impact of enzyme replacement therapy on overall survival. It has been suggested that earlier therapy, before the onset of end organ manifestations, would be more likely to prevent further damage and therefore have the biggest effect on overall survival. There is as yet little evidence to substantiate this hypothesis however clinical trials have recently demonstrated safety and therapeutic effects of enzyme replacement in children.

So far, there are only limited data available on the clinical course of the disease and adverse events in patients, switching from one therapeutic alternative to the other. West and Lemoine (16) report clinical effects of a switch from Agalsidase beta to agalsidase alfa in 5 patients with Fabry disease due to shortage of agalsidase beta. The patients were treated with Replagal® for 44 weeks at an average.

ELIGIBILITY:
Inclusion Criteria:

* Hemizygous male or heterozygous female patients at 18 years with genetically confirmed diagnosis of Anderson-Fabry disease.
* Written informed consent
* Patient had received Fabrazyme® for at least 12 months prior to starting treatment with Replagal® in full dose (i.e. 1.0 mg/kg eow) or any reduced dose prescribed by the treating physician due to the shortage of the medication
* Patient has received or is receiving treatment commercially available Replagal® (0.2 mg/kg eow) for intravenous (IV) infusion prescribed by their treatment physician and administered in accordance with the Replagal® prescribing information.
* The switch of the medication from Fabrazyme® to Replagal® had to be taken place from September 2009 onwards at the earliest
* Patient data includes disease history, measures of Fabry related disease and safety measures

Exclusion Criteria:

* Concomitant use of Fabrazyme®
* Any switch of medication from Fabrazyme® to Replagal® before September 2009
* Any switch from Fabrazyme® to Replagal® for other reasons than Fabrazyme® shortage
* Patient has received treatment with any investigational drug or device within the 30 days prior to study entry
* No written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemizygous male or heterozygous female patients at 18 years with genetically confirmed diagnosis of Anderson-Fabry disease
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Efficacy and Safety of Switch Between Agalsidase Beta to Agalsidase Alfa for Enzyme Replacement in Patients With Anderson-Fabry Disease | 24 month

CONTACTS AND LOCATIONS:
Overall Officials: Arndt Rolfs, MD, Principal Investigator
Locations (9):
- Argentina (2):
  - Juan Fernandez Hospital, Department of Neurology, Buenos Aires
  - Unidad Renal Corrientes SRL, Medicina Interna Nefrólogo, Corrientes
- UZA - University Ziekenhuis Antwerpen), Edegem, Belgium
- University Hospital "Sestre Milosrdnice" Department of neuroimmunology and neurogenetic, Zagreb, Croatia
- Miroslava Hajkova, 2nd Dept of Cardiology&Angiology, Fakultni poliklinika, Prague, Czechia
- National University Hosoital Rigshospitalet, Endokrinologisk ward, Copenhagen, Denmark
- Université de Versailles - Saint Quentin en YvelinesService de Génétique Médicale, Paris, France
- Kinderklinik München-Schwabing Städt. Klinikum GmbH, Munich, Germany
- Royal Free Hospital, Dep. of Academic Haematology, Lysosomal Storage Disorders Unit, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rolfs A, Bottcher T, Zschiesche M, Morris P, Winchester B, Bauer P, Walter U, Mix E, Lohr M, Harzer K, Strauss U, Pahnke J, Grossmann A, Benecke R. Prevalence of Fabry disease in patients with cryptogenic stroke: a prospective study. Lancet. 2005 Nov 19;366(9499):1794-6. doi: 10.1016/S0140-6736(05)67635-0. PMID 16298216
- [Background] Rolfs A, Martus P, Heuschmann PU, Grittner U, Holzhausen M, Tatlisumak T, Bottcher T, Fazekas F, Enzinger C, Ropele S, Schmidt R, Riess O, Norrving B; sifap1 Investigators. Protocol and methodology of the Stroke in Young Fabry Patients (sifap1) study: a prospective multicenter European study of 5,024 young stroke patients aged 18-55 years. Cerebrovasc Dis. 2011;31(3):253-62. doi: 10.1159/000322153. Epub 2010 Dec 21. PMID 21178350
- [Background] Kint JA. Fabry's disease: alpha-galactosidase deficiency. Science. 1970 Feb 27;167(3922):1268-9. doi: 10.1126/science.167.3922.1268. PMID 5411915
- [Background] Mehta A, Ricci R, Widmer U, Dehout F, Garcia de Lorenzo A, Kampmann C, Linhart A, Sunder-Plassmann G, Ries M, Beck M. Fabry disease defined: baseline clinical manifestations of 366 patients in the Fabry Outcome Survey. Eur J Clin Invest. 2004 Mar;34(3):236-42. doi: 10.1111/j.1365-2362.2004.01309.x. PMID 15025684
- [Background] MacDermot KD, Holmes A, Miners AH. Anderson-Fabry disease: clinical manifestations and impact of disease in a cohort of 98 hemizygous males. J Med Genet. 2001 Nov;38(11):750-60. doi: 10.1136/jmg.38.11.750. PMID 11694547
- [Background] Eng CM, Banikazemi M, Gordon RE, Goldman M, Phelps R, Kim L, Gass A, Winston J, Dikman S, Fallon JT, Brodie S, Stacy CB, Mehta D, Parsons R, Norton K, O'Callaghan M, Desnick RJ. A phase 1/2 clinical trial of enzyme replacement in fabry disease: pharmacokinetic, substrate clearance, and safety studies. Am J Hum Genet. 2001 Mar;68(3):711-22. doi: 10.1086/318809. Epub 2001 Feb 1. PMID 11179018
- [Background] Schiffmann R, Kopp JB, Austin HA 3rd, Sabnis S, Moore DF, Weibel T, Balow JE, Brady RO. Enzyme replacement therapy in Fabry disease: a randomized controlled trial. JAMA. 2001 Jun 6;285(21):2743-9. doi: 10.1001/jama.285.21.2743. PMID 11386930
- [Background] Moore DF, Altarescu G, Herscovitch P, Schiffmann R. Enzyme replacement reverses abnormal cerebrovascular responses in Fabry disease. BMC Neurol. 2002 Jun 18;2:4. doi: 10.1186/1471-2377-2-4. PMID 12079501
- [Background] Schiffmann R, Floeter MK, Dambrosia JM, Gupta S, Moore DF, Sharabi Y, Khurana RK, Brady RO. Enzyme replacement therapy improves peripheral nerve and sweat function in Fabry disease. Muscle Nerve. 2003 Dec;28(6):703-10. doi: 10.1002/mus.10497. PMID 14639584
- [Background] Hoffmann B, Reinhardt D, Koletzko B. Effect of enzyme-replacement therapy on gastrointestinal symptoms in Fabry disease. Eur J Gastroenterol Hepatol. 2004 Oct;16(10):1067-9. doi: 10.1097/00042737-200410000-00020. PMID 15371935
- [Background] Hajioff D, Goodwin S, Quiney R, Zuckerman J, MacDermot KD, Mehta A. Hearing improvement in patients with Fabry disease treated with agalsidase alfa. Acta Paediatr Suppl. 2003 Dec;92(443):28-30; discussion 27. doi: 10.1111/j.1651-2227.2003.tb00217.x. PMID 14989462
- [Background] Hoffmann B, Garcia de Lorenzo A, Mehta A, Beck M, Widmer U, Ricci R; FOS European Investigators. Effects of enzyme replacement therapy on pain and health related quality of life in patients with Fabry disease: data from FOS (Fabry Outcome Survey). J Med Genet. 2005 Mar;42(3):247-52. doi: 10.1136/jmg.2004.025791. PMID 15744039
- [Background] Beck M, Ricci R, Widmer U, Dehout F, de Lorenzo AG, Kampmann C, Linhart A, Sunder-Plassmann G, Houge G, Ramaswami U, Gal A, Mehta A. Fabry disease: overall effects of agalsidase alfa treatment. Eur J Clin Invest. 2004 Dec;34(12):838-44. doi: 10.1111/j.1365-2362.2004.01424.x. PMID 15606727
- [Background] Banikazemi M, Ullman T, Desnick RJ. Gastrointestinal manifestations of Fabry disease: clinical response to enzyme replacement therapy. Mol Genet Metab. 2005 Aug;85(4):255-9. doi: 10.1016/j.ymgme.2005.04.009. PMID 15939645
- [Background] Banikazemi M, Bultas J, Waldek S, Wilcox WR, Whitley CB, McDonald M, Finkel R, Packman S, Bichet DG, Warnock DG, Desnick RJ; Fabry Disease Clinical Trial Study Group. Agalsidase-beta therapy for advanced Fabry disease: a randomized trial. Ann Intern Med. 2007 Jan 16;146(2):77-86. doi: 10.7326/0003-4819-146-2-200701160-00148. Epub 2006 Dec 18. PMID 17179052
- [Background] Ramaswami U, Wendt S, Pintos-Morell G, Parini R, Whybra C, Leon Leal JA, Santus F, Beck M. Enzyme replacement therapy with agalsidase alfa in children with Fabry disease. Acta Paediatr. 2007 Jan;96(1):122-7. doi: 10.1111/j.1651-2227.2007.00029.x. PMID 17187618
- [Background] Ries M, Clarke JT, Whybra C, Timmons M, Robinson C, Schlaggar BL, Pastores G, Lien YH, Kampmann C, Brady RO, Beck M, Schiffmann R. Enzyme-replacement therapy with agalsidase alfa in children with Fabry disease. Pediatrics. 2006 Sep;118(3):924-32. doi: 10.1542/peds.2005-2895. PMID 16950982